CLINICAL TRIAL: NCT02582593
Title: Revitalize Cognition: A Proof of Concept Study Using Transcranial Near Infrared Stimulation in Older Adults
Brief Title: Revitalize Cognition: Near Infrared Stimulation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ed and Ethel Moore Alzheimer's Disease Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201400128; 6AZ15 (Other Grant/Funding Number: Ed and Ethel Moore Alzheimer's Disease Research Program); PF-IMP-1938 (Other Grant/Funding Number: PARKINSONS FOU)
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Aging
Keywords: Cognitive Aging; Neuromodulation; Low Level Light Therapy; Near Infrared Light; Neurostimulation
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: randomized, sham controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Older Adult Group NIR (Active Comparator): Transcranial Near Infrared Stimulation for cognitively normal participants who will attend a total of 6 treatment sessions over a two week period. During each session, stimulation via light emitting diode clusters will occur for a total of 60 minutes. Four light emitting diode (LED) clusters will be applied in 3 distinct configurations. There will be 20 minutes of stimulation at each of these 3 configurations. Each configuration will target 4 sites, for a total of 12 sites over the course of the 60 minute session. The power density used will be 500 milliwatts (mW) with a cumulative fluence (energy density) of 312 Joules/cm2 (26 J/cm2 applied at 12 sites). It is estimated that approximately 6 Joules/cm2 will reach the cortex with each daily treatment.
  Interventions: Device: MedX 1116 Rehab Console
- Older Adult Group - Sham (Sham Comparator): Cognitively Normal Participants in the sham control group will undergo identical procedures as the intervention group - screening, baseline testing, and LED cluster placement procedures. However, during the near infrared (NIR) session, the MedX console will not be turned on and no active stimulation will be applied.
  Interventions: Device: Sham MedX 1116 Rehab Console

INTERVENTIONS:
Device: MedX 1116 Rehab Console — This intervention makes use of transcranially applied near infrared light using light emitting diodes. Near infrared light will be applied to the scalp for a period of 1 hour at each session. A total of six session will be held.
  Other Names: Photobiomodulation; Low Level Light Therapy; Transcranial Near Infrared Stimulation
  Arms: Older Adult Group NIR
Device: Sham MedX 1116 Rehab Console — This intervention makes use of sham transcranially applied near infrared light using light emitting diodes. Light emitting diodes (but not near-infrared light) will be applied to the scalp for a period of 1 hour at each session. A total of six session will be held.
  Other Names: Placebo
  Arms: Older Adult Group - Sham

SUMMARY:
Changes in mood and cognition are common in older adulthood. Some studies have suggested that transcranial application of near-infrared (NIR) light may have enhancing effects on cognitive and mood status in young adults and individuals with traumatic brain injury. This effect has not been examined in older adults. This study will involve a randomized sham-controlled trial to learn whether NIR stimulation improves cognition and mood in older adults, relative to sham treated controls.

Aim 4 of this study (Parkinson Specific) is registered separately under NCT06688357

DETAILED DESCRIPTION:
There is a dearth of clinically meaningful treatment options at this point in time for individuals who are at increased risk for transitioning to dementia, particularly those with the amnestic variant of mild cognitive impairment (aMCI). While waiting for causative cures and preventive approaches, investigators are faced with the task of identifying modifying therapies that might alter the course or slow down the transition from normal cognition to MCI to dementia.

The proposed study hopes to contribute to this mission by testing the viability of a different type of intervention, one involving transcranial delivery of near-infrared (NIR) wavelengths (808-904nm). Near-infrared stimulation is safe, non-invasive and appears to improve mitochondrial function by promoting increased production of intracellular adenosine triphosphate (ATP) and possibly improved blood flow. Perhaps most compelling are recent findings of reduced beta-amyloid and neurofibrillary tangles in transgenic Alzheimer's mouse models after exposure to real vs sham transcranial NIR stimulation. Preliminary human involving traumatic brain injury (TBI), stroke, and young adult populations have also been promising in terms of positive effects of NIR on cognition.

The overall goal of the present study is to learn whether this unconventional NIR stimulation approach has potential for improving cognition in older adults. To do so, investigators will conduct a randomized sham controlled pilot trial. The intervention will involve six sessions, over a 2-week period in which real or sham stimulation is transcranially applied using a delivery system that has been FDA-approved as a nonsignificant risk since 2003. Researchers hope to learn whether NIR stimulation, relative to sham, has positive effects on cognition and mood in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 62 years or above
* Able to provide informed consent and perform cognitive and mood measures on a computer
* Willingness to be randomized to Sham or Real intervention
* Can devote 2 weeks to the intervention, and additional time for pre and post testing
* 8th grade education and ability to read on 8th grade level based on scores on the Wechsler Test of Adult Reading (WTAR) or the Wide Range Achievement Test-IV (WRAT-IV); or a reading test at 14 pt. text
* On stable doses of major medications; Since some older adults with memory complaints may be prescribed acetylcholinererase inhibitors or related medications by their primary care physicians (i.e., donepezil, rivastigmine, galantaominhe, memantime, or other potential memory-enhancing agent(s), we will not exclude them as long as they have been on stable medications for at least two months and plan to continue this medication during study participation.
* Willingness to allow a study partner (spouse, family member, friend) to answer questions about their cognitive, mood, and other behaviors

Exclusion criteria

* Sensory loss (vision, hearing) or motor deficits that would preclude participation in the experimental cognitive tasks or neuropsychological assessment
* Unstable and uncontrolled medical conditions (metabolic encephalopathy, HIV, moderate to severe kidney or liver disease)
* Previous major strokes or other known significant brain abnormalities or diseases affecting cognition (i.e., multiple sclerosis, seizure disorder, brain surgery, moderate TBI, etc.). No history of brain surgery. Exceptions are a diagnosis of Parkinson's disease for the PD subgroup.
* Evidence of potential dementia (e.g., scores < 24 on the Mini Mental State Exam (MMSE), or < 20 on the Montreal Cognitive Assessement (MoCA), or less than 5th percentile on the Dementia Rating Scale-2 (DRS-2)
* Current or past history of major psychiatric disturbance including schizophrenia, or active psychosis, bipolar disorder, current major depressive episode, current alcohol or substance abuse or history thereof within the past six months. This will be assessed using the Mental Health Screen v.3 (Carroll & McGinley), a modification of the Structured Clinical Interview for DSM-IV psychiatric disorders. We are not excluding individuals who are taking antidepressants or anti-anxiety medications, however, use of antidepressants and anxiolytics will be recorded and data will be analyzed in post-hoc analyses
* Use of antipsychotics, sedatives, or other medications with significant anticholinergic properties (due to potential influence on memory)
* Use of photo-sensitive medications such as steroids or retin-A within 15 days of the study intervention
* Diagnosis of cancer
* Previous participation in a cognitive training study within the last 3 months or current involvement in another study at VITAL or ReVITALIZE, or another study involving cognitive training or intervention at the time of participation

Ages: 62 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Bowers, Ph.D., Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - The Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - The Village Retirement Community, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The older adult cohort was recruited from the community via advertisements. Recruitment began in 2015 and ended in 2018.
  This protocol also includes participants with Parkinson disease reported in NCT-TBD.
Pre-assignment Details: Three participants dropped out prior to beginning the sham intervention due study demands and family health issues.
Groups:
- Older Adults Active Comparator NIR: In this group, participants underwent six sessions of active NIR intervention that were given over two weeks (3 sessions/week).
- Older Adult Sham Comparator NIR: Participants assigned to this group underwent six sessions of sham intervention that were given over two weeks (3 sessions/week).
Period: Overall Study
Arm/Group | Older Adults Active Comparator NIR | Older Adult Sham Comparator NIR
Started | 8 | 5 (Of the 8 individuals randomized to this intervention, 3 dropped out prior to starting the intervention or completing the baseline due to family illness and time demands)
Completed | 8 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 3 participants from the Sham Group opted not to undergo the intervention after passing screeing due to time demands and family health reasons.
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (8.1) | 74.4 (4.6) | 74.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
MoCA [Mean (Standard Deviation); unit: units on a scale] — A cognitive screening measure, the Montreal Cognitive Assessment (MoCA), was obtained on participants during the screening-baseline phase. Scores on the MoCA scale range from a minimum of 0 to maximum of 30. Higher scores mean better cognition.
  units on a scale | 28.1 (1.1) | 28.3 (1.0) | 28.2 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: NIH Examiner Battery, Executive Composite Changes From Baseline to Post-testing
Description: Computer-based battery of executive functioning tests which yields a total or "composite" score to represent global executive functioning. Executive composite scores can range from -3.0 to 3.0, with higher scores corresponding to better executive functioning, and negative scores indicating impairment. A change score will be calculated by subtracting the baseline scores from the post-test scores.
Time Frame: Change in baseline to approximately week 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham
Number analyzed (Participants) | 8 | 5
z-score | 0.33 (.5) | 0.22 (.1)
Statistical Analysis 1: Comparison: Older Adult Group NIR vs Older Adult Group - Sham; An independent sample t-test was used to examine difference in Pre-post intervention change scores for the Active and Sham groups;. Cohen's d was calculated to determine effect size; Test type: Superiority; p = .575, t-test, 2 sided — t = .581, only 1 comparison (2 groups) and thus multiple comparison correction not needed; Cohen's D = 0.27

2. Secondary Outcome: Composite Learning-Retention Score From ARENA Task
Description: ARENA is a task of spatial memory and navigation that is a human analogue to the Morris water maze used in animal studies. Participants learn to navigate to a hidden target location relying on spatial cues in a simulated environment over a series of 8 learning trials and a final retention trial. The final ARENA outcome is an Overall Composite z-score combining learning and retention metrics as follows: [-Learning z-score + Retention z-score]/2. The learning z-score is based on two metrics (path length to target, time to reach target) that are converted to z-scores and averaged over the 8 learning trials. The retention z-score is based on percent time spent in the target quadrant during the retention trial. The Learning and Retention z-scores are combined to create a single final Arena Composite outcome. Higher composite scores reflect better memory performance. A change score is calculated by subtracting the Baseline Composite score from the post-test Composite Score
Time Frame: Change in baseline to approximately week 3
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham
Number analyzed (Participants) | 8 | 5
z-score | 0.17 (.6) | -.41 (.5)
Statistical Analysis 1: Comparison: Older Adult Group NIR vs Older Adult Group - Sham; independent t-test, cohen's d effect size; Test type: Superiority; p = .160, t-test, 2 sided — t = 1.574; only two comparisons, thus not necessary to adjust; Cohen's D = 1.06

3. Secondary Outcome: NIH Toolbox Emotion Psychological Wellbeing Scale Changes From Baseline to Post-testing
Description: The Psychological Wellbeing Scale from the NIH Toolbox Emotion module Wellbeing Scale results in T-scores (mean=50, SD=10) for categories such as positive affect, life satisfaction, and meaning and purpose. Scores below 40 indicate low levels of wellbeing and scores above 60 indicating high levels of wellbeing. Change scores will be calculated by subtracting the baseline scores from the post-test scores.
Time Frame: Change in baseline to approximately week 3 (Post - Baseline)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham
Number analyzed (Participants) | 8 | 5
T-score | -0.04 (7.8) | -3.50 (5.3)
Statistical Analysis 1: Comparison: Older Adult Group NIR vs Older Adult Group - Sham; independent t-test, Cohen's d effect size; Test type: Superiority; p = .424, t-test, 2 sided; Cohen's D = 0.27

4. Secondary Outcome: NIH Toolbox Emotion Negative Affect Scale Changes From Baseline to Post-testing
Description: The Negative Affect Scale from the NIH Toolbox Emotion module results in T-scores (mean=50, SD=10) for categories such as anger, sadness, and apathy. Scores below 40 indicate low levels of negative affect and scores above 60 indicate high levels of negative affect. Change scores will be calculated by subtracting the baseline scores from the post-test scores.
Time Frame: Change from baseline to approximately week 3 (Post Intervention - Baseline)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham
Number analyzed (Participants) | 8 | 5
T-score | -1.92 (3.6) | 2.11 (4.5)
Statistical Analysis 1: Comparison: Older Adult Group NIR vs Older Adult Group - Sham; independent sample t-test, Cohen's d effect size; Test type: Superiority; p = 0.099, t-test, 2 sided — no adjustment necessary, only 1 comparison; Cohen's D = -1.03

ADVERSE EVENTS:
Time Frame: 3 weeks; collected during intervention and during post-evaluation
Description: Does not differ
Arm/Group | Older Adult Group NIR | Older Adult Group - Sham
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5

LIMITATIONS AND CAVEATS:
This was pilot proof of concept study designed to determine potential effect sizes for a larger study. Small sample size was major limitation. Instead of using overall executive composite score as from the NIH Examiner as major outcome, we recommend breaking down executive function into its components (working memory, fluency) in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02582593/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT02582593/SAP_001.pdf